CLINICAL TRIAL: NCT00799019
Title: A Prospective, Immunogenicity Surveillance Registry of Erythropoiesis Stimulating Agent (ESA) With Subcutaneous Exposure in Thailand
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, Kearkiat Praditpornsilpa, Associated Professor, Chulalongkorn University
Other Study IDs: MDCU 1/2008; IRB No.404/50; Ref. No.2/2551
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Erythropoietin
Keywords: EPO antibody mediated PRCA; Erythropoiesis stimulating agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This multicenter, immunogenicity surveillance registry employs a prospective, cohort design for patients who are using erythropoiesis stimulating agents (ESA)according to normal practice consistent with the medical indications. Subjects will be observed for the development of immunogenicity and PRCA for up to 3 years. Information on exposure to ESA products, ESA product handling and storage, and most recent hemoglobin level will be collected quarterly in the case report form. For cases of suspected PRCA, that sera specimen will be tested for EPO antibodies at Division of Nephrology, Chulalongkorn University Laboratory.

An Advisory Board (ADB) will periodically review blinded case data for subjects with unexplained loss of efficacy (LOE), identify cases of EPO antibody-mediated PRCA and will be responsible for data summary and make recommendations related to the incidence rate of PRCA associated with S.C. ESA use. The registry will provide no inducement to change therapy and will be non-interventional. The primary objective for this study is to estimate the incidence of anti-human Erythropoiesis and anti-EPO PRCA, develop in such patients. The diagnosis of PRCA by bone marrow biopsy must be prerequisite before the antibody assay. The secondary objective is to evaluate the efficacy of ESA for treatment of erythropoiesis deficiency anemia. Registry subjects will be adult men and women who are receiving or about to receive (within 1 month) a marketed ESA product by the s.c. route of administration at the time of enrollment. The marketed ESAs include innovative ESA and biosimilar ESA. Potential subjects will only be enrolled if they have been receiving an Erythropoiesis product for less than 1 year. Cases of EPO antibody-mediated PRCA will be determined by the clinical presence of essential criteria of unexplained LOE, administration of ESA product, bone marrow biopsy diagnosis of PRCA, and presence of EPO antibody. The sera of patients who meet all criteria will be assayed for neutralization.

DETAILED DESCRIPTION:
Incidence rates of EPO antibody-mediated PRCA will be estimated as the total number of cases of anti-Erythropoiesis and anti-EPO antibodies mediated PRCA attributed to a specific product presentation divided by the person-year (PY) of s.c. exposure. Incidence rates will be adjusted for duration of exposure by stratification. Sensitivity analyses with varying assumptions on the latency from exposure with Erythropoiesis product to onset of PRCA will be employed in general and will be evaluated specifically if subjects switch therapy, have mixed exposure to multiple ESA products by the s.c. route of administration, or discontinue therapy and remain under observation. Confidence intervals for rate estimates will be calculated using the Poisson distribution for rare events.

ELIGIBILITY:
Inclusion Criteria:

* Be receiving or about to receive (within 1 month) a marketed erythropoiesis product by the s.c. route of administration
* Be 18 years of age or older
* Be likely to continue to receive s.c. erythropoiesis product(s) for at least 1 year
* Have read and signed the informed consent document for this registry indicating that they understand the purpose of and procedures required for the registry and are willing to participate in the registry.

Exclusion Criteria:

Potential subjects who meet any of the following criteria are excluded from the registry:

* Inability of the treating physician to obtain adequate follow-up information
* Have a history of PRCA or aplastic anemia
* Are experiencing unexplained loss or lack of effect (LOE) to a recombinant erythropoiesis product ongoing at the time of enrollment
* Have had prior recombinant erythropoiesis treatment whose anemia had never responded (primary lack of efficacy)
* Have a history of EPO antibodies prior to enrollment
* Are currently receiving immunosuppressive medication (e.g., cyclosporine, tacrolimus, sirolimus, mycophenolic mofetil, azathioprine, or monoclonal antibodies) and prednisolone.
* Have previously participated in this registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registry subjects will be adult men and women who are receiving or about to receive (within 1 month) a marketed ESA product by the s.c. route of administration at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2008-07; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Positive anti-erythropoietin antibody | within 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Kearkiat Praditpornsilpa, MD, Principal Investigator — Chulalongkorn University